CLINICAL TRIAL: NCT07029048
Title: Longitudinal Evaluation of Oxidative Stress Biomarkers and Cognitive Impairment in Post-COVID-19 Patients: A Prospective Observational Study
Brief Title: Oxidative Stress and Cognitive Dysfunction After COVID-19
Status: Completed | Type: Observational
Sponsor: Karaganda Medical University (Other)
Responsible Party: Principal Investigator, Yessenbay Gulfairuz, Principal Investigator Zhumabekova Indira, Karaganda Medical University
Other Study IDs: OXYSTRESS-COVID-19
Record Dates: First submitted 2025-06-17; First posted 2025-06-19 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: COVID 19; Oxydative Stress; Cognitive Impairments
Keywords: COVID 19; cell-free DNA; Neutrophil Extracellular Trap; AOPP; memory; attention
MeSH Terms: conditions — COVID-19; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-COVID-19 survivors followed over 12 months: Primary Objective:
  To investigate the association between oxidative stress biomarkers (e.g., cell-free DNA, AOPP, NETs, OMB, NO) and cognitive impairment (memory and attention deficits) in post-COVID-19 patients.
  Secondary Objectives:
  To assess the longitudinal dynamics of oxidative stress markers at 0-3, 3-6, and 6-12 months post-COVID.
  To identify biochemical predictors of persistent cognitive dysfunction.
  Interventions: Other: Standard Post-COVID Rehabilitation Program

INTERVENTIONS:
Other: Standard Post-COVID Rehabilitation Program — This standardized rehabilitation intervention includes a 14-day inpatient course comprising physiotherapy, therapeutic exercises, massage, and respiratory gymnastics. The program is delivered equally to all participants regardless of cognitive status and is intended to promote post-viral recovery in patients recently discharged following COVID-19 pneumonia. No specific cognitive therapy or pharmacological treatment is administered during the rehabilitation period. The intervention is used as background care, not as an experimental variable.

SUMMARY:
This observational cohort study will investigate the association between oxidative stress biomarkers and post-COVID-19 cognitive impairment. A total of 45 recovered COVID-19 patients aged 30-65 will be enrolled and followed at three intervals: 0-3, 3-6, and 6-12 months post-infection. Cognitive function will be assessed using standardized memory and attention tests, while venous blood samples will be analyzed for nitric oxide, AOPP, NETs, and extracellular nucleic acids. The study aims to identify early predictors of long COVID cognitive sequelae and evaluate biological mechanisms underlying persistent neurocognitive symptoms.

DETAILED DESCRIPTION:
This prospective observational cohort study will aim to investigate whether markers of oxidative stress, including advanced oxidation protein products (AOPP), nitric oxide (NO), extracellular nucleic acids (DNA/RNA), and neutrophil extracellular traps (NETs), can predict cognitive dysfunction in patients recovering from COVID-19 pneumonia.

Post-viral cognitive impairment, commonly referred to as "brain fog," has emerged as a major complication in long COVID patients. The estimated prevalence of neurocognitive deficits ranges from 21% to 65% depending on disease severity and follow-up duration . Even individuals with mild infection can present with persistent impairments in memory, attention, and executive function .

Growing evidence suggests that oxidative stress plays a critical role in neurodegeneration and long-COVID symptoms . SARS-CoV-2 triggers an "oxidative storm," marked by excess production of reactive oxygen and nitrogen species, causing cellular injury . These species impair neurovascular coupling and lead to persistent endothelial dysfunction and neuroinflammation . Furthermore, cell-free DNA and RNA, key damage-associated molecular patterns (DAMPs), act as immune triggers via Toll-like receptor pathways .

Another mechanism under scrutiny is NETosis, the extrusion of web-like neutrophil traps that damage endothelial cells, increase blood-brain barrier permeability, and drive systemic inflammation . Elevated NETs have been found in acute and chronic COVID-19 cases and may be a biomarker of persistent inflammation and thrombosis .

Despite the biological plausibility of these mechanisms, there is limited longitudinal human data linking oxidative stress markers to cognitive outcomes in COVID-19 survivors. This study will follow participants for one year, evaluating neurocognitive performance and biochemical markers at three post-infection intervals: 0-3, 3-6, and 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Confirmed history of COVID-19 pneumonia (PCR and CT-verified)
* Recovered and discharged from COVID-19 hospital unit
* Able to provide informed consent
* Either presence or absence of self-reported cognitive complaints

Exclusion Criteria:

* History of CNS disease (e.g., dementia, stroke, TBI)
* Psychiatric illness
* Decompensated comorbidities (diabetes, cardiovascular, renal, or hepatic failure)
* Alcohol/drug abuse
* Uncontrolled hypertension
* Acute respiratory insufficiency or fever at time of assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will involve adult patients who have recovered from PCR-confirmed COVID-19 pneumonia. Participants will be recruited at the time of discharge from inpatient treatment facilities in Karaganda, Kazakhstan. The target population includes individuals with or without subjective cognitive complaints during early recovery. All participants must have preserved consciousness at baseline, be able to provide informed consent, and meet the inclusion and exclusion criteria related to neuropsychiatric, respiratory, and systemic comorbidities. A balanced representation of genders will be encouraged. The study will longitudinally assess cognitive and biochemical parameters at three post-infection intervals: 0-3 months, 3-6 months, and 6-12 months.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Wechsler Memory Scale (WMS) Scores | Measured at 0-3, 3-6, and 6-12 months after discharge.
  Assessment of memory function using the Wechsler Memory Scale, which measures different memory domains including working memory, visual memory, and auditory memory.
  Scoring Range: 50 to 150 (higher scores indicate better memory performance).
Change in Bourdon Attention Test Scores | Measured at 0-3, 3-6, and 6-12 months after discharge.
  Assessment of sustained attention and processing speed using the Bourdon Attention Test, which records the number of correctly marked target symbols within a given time.
  Scoring Range: 0 to 15 (higher scores indicate better attention and processing accuracy).

SECONDARY OUTCOMES:
Levels of Nitric Oxide (NO), AOPP, and Oxidised Proteins | Measured at 0-3, 3-6, and 6-12 months after discharge.
  Measured via blood analysis at three time points.
Extracellular DNA/RNA and CRF nucleic acids | Measured at 0-3, 3-6, and 6-12 months after discharge.
  Quantified in plasma and erythrocytes.
Neutrophil Extracellular Trap (NET) Levels | Measured at 0-3, 3-6, and 6-12 months after discharge.
  Expressed as % of neutrophils, visualised microscopically.

CONTACTS AND LOCATIONS:
Locations (1):
- Karaganda Medical University, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1. Premraj L, Kannapadi NV, Briggs J, Seal SM, Battaglini D, Fanning J, et al. Mid and long-term neurological and neuropsychiatric manifestations of post-COVID-19 syndrome: A meta-analysis. J Neurol Sci. 2022;434:120162. 2. Becker JH, Lin JJ, Doernberg M, Stone K, Navis A, Festa JR, et al. Assessment of Cognitive Function in Patients After COVID-19 Infection. JAMA Netw Open. 2021;4(10):e2130645. 3. Graham EL, Clark JR, Orban ZS, Lim PH, Szymanski AL, Taylor C, et al. Persistent neurologic symptoms and cognitive dysfunction in non-hospitalized Covid-19 "long haulers". Ann Clin Transl Neurol. 2021;8(5):1073-1085. 4. Taquet M, Geddes JR, Husain M, Luciano S, Harrison PJ. 6-month neurological and psychiatric outcomes in 236,379 survivors of COVID-19. Lancet Psychiatry. 2021;8(5):416-427. 5. Hosp JA, Dressing A, Blazhenets G, Bormann T, Rau A, Schwabenland M, et al. Cognitive impairment and altered cerebral glucose metabolism in the subacute stage of COVID-19. Brain. 2021;144(4):1263-1276. 6. Cichoż-Lach H, Michalak A. Oxidative stress as a crucial factor in liver diseases. World J Gastroenterol. 2014;20(25):8082-8091. 7. Delgado-Roche L, Mesta F. Oxidative Stress as Key Player in Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV) Infection. Arch Med Res. 2020;51(5):384-387. 8. Cecchini R, Cecchini AL. SARS-CoV-2 infection pathogenesis is related to oxidative stress as a response to aggression. Med Hypotheses. 2020;143:110102. 9. Islam MT, Sarkar C, El-Kersh DM, Jain S, Mitra S, Debnath M, et al. COVID-19 and neurodegeneration: The contribution of oxidative stress and inflammation. Oxid Med Cell Longev. 2022;2022:9503143. 10. Cheignon C, Tomas M, Bonnefont-Rousselot D, Faller P, Hureau C, Collin F. Oxidative stress and the amyloid beta peptide in Alzheimer's disease. Redox Biol. 2018;14:450-464. 11. Maes M, Vojdani A, Galecki P. Redox dysregulation, immuno-inflammatory pathways, and neuropsychiatric disorders in Long COVID. Mol Neurobiol. 2022;59(3):1859-1882.